CLINICAL TRIAL: NCT05528640
Title: The Effectiveness of an Educational Program on the Mental Health Literacy of Nurses Working in General Hospitals: a Controlled Trial
Brief Title: Interventional Study of Mental Health Literacy Educational Program for General Hospital Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHEUNG, Janice, Student, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1155149877
Record Dates: First submitted 2022-06-01; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Mental Health Issue
Keywords: Education; Mental health literacy; Nurses; General hospital

STUDY DESIGN:
Intervention Model Description: This study is a prospective 2-arm parallel controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health Literacy Educational Program (Experimental): An educational program consisting of six 30-minutes online educational sessions and one 60-minutes face-to-face session.
  Interventions: Other: Mental Health Literacy Program
- Control Group (No Intervention): No active intervention

INTERVENTIONS:
Other: Mental Health Literacy Program — Six educational sessions will be delivered on a private YouTube channel which consists of information about mental health literacy (knowledge about priority mental illnesses, attitude/ stigma related to mental illnesses, and help-seeking efficacy). There will be six-weeks unrestricted access period. Afterwards, the round-up session which consists of problem-based learning and group sharing will be delivered in person. Two vignettes based on the clinical scenarios will be given for discussion. Furthermore, participants are encouraged to share their opinion on mental health literacy, strategies for dealing with difficulties of caring for patients with mental illnesses in general hospitals, way to promote mental health literacy of healthcare professionals in general hospitals
  Arms: Mental Health Literacy Educational Program

SUMMARY:
Mental health literacy is a concept that encompasses knowledge of mental health, mental illnesses, and their management; mental illness-related attitudes/ stigma; and help-seeking efficacy. It impacted care provision by affecting healthcare professionals' ability to recognize, manage and prevent mental illnesses. It was found that physical-mental comorbidity (co-occurrence of physical and mental illnesses) imposed a burden on patients and the healthcare system. However, the referral rate to psychiatric consultation-liaison in general hospitals was low could be attributed to the suboptimal level of mental health literacy of general hospital healthcare professionals. Nurses are the major healthcare workforce in general hospitals for the initial identification of mental illness, help doctors to deal with patients' conditions, and make a contribution to positive patient outcomes in general hospitals. Therefore, there is an urgent need to improve the mental health literacy of nurses working in general hospitals.

An education program had been developed guided by the concept of mental health literacy, and self-efficacy theory. This study aims to examine the effect of an educational program on improving the mental health literacy of general hospital nurses, in terms of knowledge of mental health, mental illnesses, and their treatment; attitude or stigma about mental illnesses; and help-seeking efficacy. It also measures the interventional effect on perceived competency in caring for patients with mental illness and work stress among general hospital nurses, as well as patient satisfaction with nursing care in general hospitals.

DETAILED DESCRIPTION:
This study is a prospective 2-arm parallel controlled trial. The study sites will be conducted in the emergency departments and medical wards of two similar regional general hospitals. It is estimated using GPower that a sample size of 64 participants per group is adequate to detect an effect size of 0.5 on the primary outcomes at a post-intervention time point with 80% power at a 5% level of significance. Participants will be assigned to either an intervention group or a control group. Participants in the intervention group will receive a Mental Health Literacy Program consisting of six 30-minutes online educational sessions and one 60-minutes face-to-face session. No active intervention will be given to the control group. Outcome measures will be measured by the Mental Health Literacy Scale, the Behavioral Health Care Competency survey, the Workplace Stress Scale, and Hospital Patient Satisfaction Survey at baseline, immediately after intervention, and one-month after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Full-time registered nurse (general) or enrolled nurse (general)
* Take care for adult patients in emergency departments or medical ward

Exclusion Criteria:

* Does not understand Chinese and English
* Unable to access or use the internet.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-01-18 (Estimated); Study Completion 2023-04-21 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in level of mental health literacy | Baseline, immediately after intervention, one month after intervention
  The level of participant's mental health literacy will be evaluated using The Mental Health Literacy Scale developed by Connor & Casey (2015). This questionnaire comprised 35 items which consisted of the ability to recognize disorders (8 questions), knowledge of where to seek information (4 questions), knowledge of risk factors and causes (2 questions), knowledge of self-treatment (2 questions), knowledge of professional help available (3 questions), attitudes that promote recognition or appropriate help-seeking behavior (16 questions) (O'Connor & Casey, 2015). Questions with a 4-point scale are rated "1" was very unlikely/unhelpful, "4" was very likely/helpful and for a 5-point scale that "1" strongly disagreed/definitely unwilling, "5" strongly agreed/definitely willing. The higher the total score indicates a higher level of mental health literacy.

SECONDARY OUTCOMES:
Change from baseline in perceived competency in caring for patients with mental illnesses | Baseline, immediately after intervention, one month after intervention
  The Behavioral Health Care Competency survey will be used to assess the perceived competency in caring for patients with mental illnesses. It consists of 23-items to assess the participants' perception of their competency in assessment, intervention, recognition of the need for referral, and dealing with resources issues (Rutledge et al., 2013; Rutledge et al., 2012). Questions with a 5-point Likert-type scale with responses 1= "Strongly disagree" to 5=" Strongly agree" The higher the total score, the higher respondent's perceived competency in caring for patients with mental illnesses.
Change from baseline in level of work stress | Baseline, immediately after intervention, one month after intervention
  The Workplace Stress Scale developed by the Marlin Company will be used to assess participants' work stress levels. This scale consists of eight items that describe the perception of the respondent toward his or her work. Questions with a 5-point scale are rated "1' was never, and "5" was very often. The higher the total score indicates a higher level of work stress. A total score of 15 or lower interpreted as stress is not much of an issue, whilst 31-40 was indicative of a potentially dangerous stress level that may need to seek professional assistance.
Change from baseline in patient satisfaction with nursing care | Baseline, immediately after intervention, one month after intervention
  Hospital Patient Satisfaction Survey will be used to assess the patient satisfaction with nursing care in general hospitals. There are eight questions on the scale to measure patient satisfaction with nursing care during the hospitalization with a 4-point Likert scale (from "0"=never to "4"=always).

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT05528640/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT05528640/ICF_001.pdf